CLINICAL TRIAL: NCT01389492
Title: Nutritional Study:The Effect of Meat and Food Drived Polyphenols on Oxidize LDL Level
Brief Title: The Effect of Meat and Food Drived Polyphenols on Oxidize LDL Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Daniel Schurr, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MWPP09-HMO-CTIL
Record Dates: First submitted 2011-07-03; First posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: meat; LDL; MDA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- frozen meat (Other): 250 g of frozen meat meal for 4 days
  Interventions: Other: frozen meat cutlets meal; Other: meat meals
- frozen meat and wine (Other): 250 g of frozen meat and red wine for 4 days
  Interventions: Other: frozen meat cutlets meal; Other: meat meals
- fresh meat (Other): 250 g of fresh meat meal
  Interventions: Other: frozen meat cutlets meal; Other: meat meals
- fresh meat and wine (Other): 250 g of fresh meat meal
  Interventions: Other: frozen meat cutlets meal; Other: meat meals

INTERVENTIONS:
Other: frozen meat cutlets meal — 250 g of meat cutlets
Other: meat meals — 250 g of meat meal for 4 days

SUMMARY:
The postprandial increase in MDA level following meat meal could cause modification to LDL particles in healthy volunteers. Co-consumption of food drived polyphenols with the meat will result in a significant decrease in LDL modification.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, normal BMI

Exclusion Criteria:

* Metabolic disorders
* Smokers
* Drinkers
* Taking nutritional supplement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in plasma MDA levels following meat meal | Fasting before meal and 3, and 6 h postprandial, and fasting levels
  After an overnight fast baseline (0 h) fasting blood sample (10 ml) was collected in EDTA-treated tubes. The subjects then ate a test meal within 30 min. Blood samples (10 ml) were drawn 3 and 6 h after the meal was eaten. Serum was separated from whole blood by centrifugation (910 g, 15 min), and MDA was evaluated by HPLC in plasma samples
Changes in MDA concentration on LDL fraction following meat meals | Fasting, before meal was eaten, 3 h following meal, at day 4, 3 h following meal consumption, and day 5 following over nigth fast
  Subject consumed the test meals for 4 days. Day 1, (0 h) fasting blood sample (10 ml) was collected in EDTA-treated tubes. The sbjects then ate a test meal within 30 min. Blood samples (10 ml) were drawn 3 h after the meal was eaten. Blood was collected at day 4, 3 h after the meal was eaten, at the morning of day 5.Plasma LDL was isolated using a single discontinuous density gradient ultracentrifugation. The protein concentration was determined based on the method of Bradford. MDA concentration was evaluated by HPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Gorelik, PhD, Study Director — Hebrew University of Jerusalem
Locations (1):
- The Hebrew University of Jerusalem, Jerusalem, Israel